CLINICAL TRIAL: NCT02088632
Title: A Randomized, Double-Blind, Placebo-Controlled, Add-on Therapy Study of Xeomin (Incobotulinumtoxina) Versus Placebo in the Treatment of Trigeminal Neuralgia
Brief Title: Incobotulinum Toxin for the Treatment of Trigeminal Neuralgia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enrolled in a timely manner.
Sponsor: Thomas Jefferson University (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XEO/SDS/01
Record Dates: First submitted 2014-03-04; First posted 2014-03-17 (Estimated); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — incobotulinumtoxinA; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Incobotulinumtoxina (Active Comparator): Xeomin 25-100 units injected to chosen area one time.
  Interventions: Biological: Incobotulinumtoxina
- Placebo Comparator (Placebo Comparator): Placebo Comparator is 1-2 ml normal saline solution injected to chosen area one time.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Biological: Incobotulinumtoxina — Incobotulinumtoxina (Xeomin) is botulinum toxin type A and is administered via intramuscular injection.
  Other Names: Xeomin
  Arms: Incobotulinumtoxina
Other: Placebo Comparator — Normal saline is sterile sodium chloride without and preservatives.
  Other Names: Normal Saline, sodium chloride, placebo
  Arms: Placebo Comparator

SUMMARY:
IncobotulinumtoxinA (Xeomin®) is a neurotoxin which inhibits the release of certain chemicals at the nerve terminals. It blocks cholinergic transmission at the neuromuscular junction by inhibiting the release of acetylcholine from motor neurons. In addition it blocks the release of Substance P (SP) and Calcitonin Gene Related Peptide (CGRP) from C fibers involved in pain perception. This study is designed to see if Xeomin® is superior to placebo in the treatment of medically refractory trigeminal neuralgia (TN). Subjects will be asked to maintain an attack diary throughout the study. They will also be asked to attend 4 office visits; Visit 1- Screening Visit, Visit 2- Injection Visit, Visit 3- Follow-Up Visit and Visit 4- Final Visit. At the end of the study the active (Xeomin®) and placebo groups will be compared to see if one group had better relief than the other.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, add-on therapy study. Up to 70 eligible subjects with medically refractory TN will be screened to enroll forty subjects; twenty will be randomized to the active medication group IncobotulinumtoxinA (Xeomin) and twenty to the placebo group (0.9% Normal Saline Solution). Using a daily diary, all subjects will document their overall pain level and attack frequency and intensity for four weeks. After the four week baseline period, subjects will undergo initial injections (IncobotulinumtoxinA [Xeomin] or placebo). Subjects will remain on a consistent dose of their previously prescribed medications throughout the study.

The primary outcome will be the difference in decrease in mean number of attacks of at least 4/10 intensity between the active and placebo groups. Secondary outcome measures will be frequency and average intensity of daily pain attacks. Subject Global Assessment, Beck Depression Inventory II (BDI-II), Short Form-36 (SF-36) Health Surveys, and visual analog scale (VAS), will also be assessed.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria

* Age 18 - 75 yrs
* Male or non-pregnant/non-lactating female
* Subjects must have a mean attack frequency of at least 3 episodes/day of 4/10 pain
* Use of adequate birth-control measures as determined by investigator for females of child-bearing potential
* Diagnosis of Classical trigeminal neuralgia (TN) using International Classification of Headache Disorders (ICHD-2) criteria (see Appendix A in Protocol)
* Subjects have given written informed consent prior to entering study
* Subjects on a stable dose of concomitant preventive medications for treatment of TN for at least 4 weeks prior to study entry and throughout the 12 week observation period
* Subjects who require "rescue" analgesic medication during the study will be allowed to use their current (pre-study) opioid and/or non opioid analgesics as clinically indicated (e.g., non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen, cyclooxygenase-2 (COX-2) inhibitors, topical analgesics).
* Subjects will be prohibited from initiating any therapy with a new preventive medication throughout the remainder of the study.
* Subject must be willing and able to abstain from initiating an alternative therapy (e.g., acupuncture, massage or physical therapy) for pain relief during the study.

(NOTE: subjects who are currently using alternative therapy for pain relief can be enrolled if they are willing and able to maintain such therapy stable throughout the study.)

-

Exclusion Criteria:Exclusion Criteria

* Symptomatic TN
* Serious hepatic, respiratory, hematologic, cardiovascular or renal condition
* Neurologic pain other than TN, with the exception of occasional migraine or tension-type headaches. (<4 headaches per month; < 10 headache days/month)
* Psychiatric or medical condition that might compromise participation in study, as determined by the investigator
* Administration of any investigational drug within 30 days prior to screening
* History of substance abuse/alcoholism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2015-06-11 (Actual); Study Completion 2016-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Silberstein, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Jefferson Headache Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The original target enrollment was 70 subjects
Pre-assignment Details: Actual enrollment was 6. Recruitment efforts were limited to patients in our practice who could come in for visits and few responded to recruitment efforts. The appointment openings/schedule for visits was very limited.
Period: Overall Study
Arm/Group | Incobotulinumtoxina | Placebo Comparator
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IncobotulinumtoxinA | Placebo Comparator | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 54.3 [42 to 68] | 49.6 [43 to 63] | 52.0 [42 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Number of Headache Attacks Reported in Active and Placebo Group
Description: Mean daily number of attacks during baseline period (30 days) will be compared to mean daily number of attacks for baseline and 84 days as recorded in patient diary.
Time Frame: 84 days
Population: Patients treated with Xeomin and patients treated with placebo
Measure: Mean (Standard Deviation); unit: attacks per day
Groups:
- Active: Received Xeomin injections
- Placebo Group: Placebo group Did not receive xeomin
Arm/Group | Active | Placebo Group
Number analyzed (Participants) | 3 | 3
attacks per day | 1.96 (2.9) | -200.133 (286.9)

2. Secondary Outcome: Change in Mean Pain Intensity of Active and Placebo Group
Description: Mean of the daily pain intensity as measured on a 0-10 pain scale where 0 = no pain and 10 is the worst pain reported on paper diary from baseline and 84 days
Time Frame: 84 days
Population: Descriptive statistics only
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active: Subjects who received Xeomin injections
- Placebo: Subjects received placebo injections
Arm/Group | Active | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | -2.66 (.98) | .73 (.54)

ADVERSE EVENTS:
Time Frame: Adverse events collection was from start of consent to end of study - approximately 84 days
Arm/Group | Incobotulinumtoxina | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incobotulinumtoxina (N=3) | Placebo Comparator (N=3)
Drowsiness (General disorders) | 1 (1) | 0 (0)
muscle weakness (General disorders) | 1 (1) | 0 (0)
Aphthous ulcers (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Numbness left temple (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Very slow enrollment and low number of participants limited study. Study was terminated prior to analysis. The data was highly skewed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No